CLINICAL TRIAL: NCT05143658
Title: Comparison of Laparoscopic Pectopexy and Laparoscopic Lateral Suspension Techniques in Uterine-preserving Apical Prolapsus Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ozan Karadeniz, Principal investigator, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KanuniSSS
Record Dates: First submitted 2021-10-28; First posted 2021-12-03 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Pelvic Organ Prolapse
Keywords: pectopexy; lateral suspension; pelvic organ prolapse; uterine sparing; laparoscopy
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Lateral Suspension Group (LLS) (Active Comparator): Anterior and apical prolapse repair via LLS
  Interventions: Procedure: LLS versus LP
- Laparoscopic Pectopexy (LP) (Experimental): Anterior and apical prolapse repair via LP
  Interventions: Procedure: LLS versus LP

INTERVENTIONS:
Procedure: LLS versus LP — Procedure: Laparoscopic repair of anterior and apical pelvic organ prolapse Surgical correction of anterior and apical pelvic organ prolapse by laparoscopy

SUMMARY:
The aim of the study will be to compare the laparoscopic pectopexy (LP) and laparoscopic lateral suspension (LLS) techniques in the management of uterine sparing apical prolapse (POP-Q >2) at 1 year and yearly up to 2 years.

DETAILED DESCRIPTION:
Primary and secondary endpoints:

Primary outcome measures will be the subjective cure of prolapse ("absence or presence of a bulge in the vagina"), objective success with anatomic absence of advanced prolapse at POP-Q sites Ba, C and Bp defined as less than 1 cm individually and as a total.

Secondary outcome measures include all other parameters such as perioperative outcomes, patient satisfaction, quality of life outcomes, complications, scores on questionnaires, and reoperations.

The study protocol will be submitted to the institutional review boards of every participating study site and written informed consent will be obtained from all participants on enrolment.

Project design: The investigators will perform an international multicentre single-blind randomized controlled trial with participating our tertiary referral hospital.

ELIGIBILITY:
Inclusion Criteria:

* Women with symptomatic stage 2 or greater (point C -1 or more pelvic organ prolapse quantification POP-Q) apical prolapse

Exclusion Criteria:

* Women not eligible for surgery for medical or anesthesiological reasons
* Inability to comprehend questionnaires
* Inability to give informed consent
* Inability to return for a review
* Prior laparoscopic prolapse repair
* Prior vaginal mesh prolapse procedure
* Severe cardiovascular or respiratory disease
* Women who don't want uterine preserving surgery
* Pregnancy
* Age <18 years, Age >45 years

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Subjective cure rate of prolapse | [ Time Frame: 12 months after intervention ]
  Provided by the patient's feeling of the "Absence of a bulge in the vagina"
Objective success | [ Time Frame: 12 months after intervention ]
  Defined as anatomic absence of advanced prolapse at POP-Q sites Ba, C and Bp defined as less than 1 cm individually and as a total

SECONDARY OUTCOMES:
Prolapse-related Quality of life | [ Time Frame: 12 months after intervention ]
  This will be assessed using a validated questionnaire (Prolapse Quality of Life questionnaire P-QoL) The questionnaire contains 9 domains. Each answer of the patient will have values that range between 1 to 4 or 1 to 5 for the 1st question only). (1 very good 4/5 very poor). There is no overall score. A symptomatic woman might have only one domain impaired and another one might have all domains impaired. We consider both of them symptomatic but in different or same aspects of quality of life. To differentiate different domains, it is important for the decision of our surgery (we will be careful in shortening and narrowing a vagina of a woman who had only a preoperative high (impaired) Personal relationships domain score and other domains in the normal range).
  This will also help us in the follow up visits.
Failure (%) | [ Time Frame: 12 months after intervention ]
  Recurrence rate
Complications | [ Time Frame: 12 months after intervention ]
  İnjury ( bowel, intestinal, blood vessel injuries, mesh erosions)
Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) | [ Time Frame: 12 months after intervention ]
  The PISQ-12 is a self-adminestered questionnaire that evaluates sexual function of women with pelvic organ prolapse or urinary incontinence. The questionnaire has 12 items. Other than the first 4 questions that are scored from 4 to 0, all questions are scored from 0 to 4. The total score is calculated with totaling the score of each question. The maximum score is 48. Higher scores show good sexual functioning of women.
Incontinence Impact Questionnaire (IIQ-7) | [ Time Frame: 12 months after intervention ]
  evaluating the impact of urinary incontinence
Pelvic Floor Distress Inventory (PFDI - 20) | [ Time Frame: 12 months after intervention ]
  evaluating the bowel, bladder, or pelvic symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ozan Karadeniz, MD, Principal Investigator — Kanuni Sultan Suleyman Training and Research Hospital
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)